CLINICAL TRIAL: NCT03711175
Title: A Prospective Multicenter Study to Examine the Influence of Repairing the Sub-scapularis on Outcomes After Reverse Arthroplasty: A Randomized, Controlled Trial.
Brief Title: The Influence of Repairing the Sub-scapularis on Outcomes After Reverse Arthroplasty
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PS-903
Record Dates: First submitted 2018-10-11; First posted 2018-10-18 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Severe Arthropathy With a Grossly Deficient Rotator Cuff
Keywords: Sub-scapularis repair

STUDY DESIGN:
Intervention Model Description: Two treatment arms. One group will have the subscapularis repaired during surgery, and one group will not have the subscapularis repaired during surgery. All subjects will receive the same device.
Who Masked: Participant
Masking Description: Subject will not know which group they were randomized to until the completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Other): The subscapularis is repaired. Receives device
  Interventions: Procedure: Subscapularis repair; Device: Shoulder implant
- Group B (Other): The subscapularis is not repaired. Receives device
  Interventions: Device: Shoulder implant

INTERVENTIONS:
Procedure: Subscapularis repair — Utilizing fiberwire, high tensile strength suture
  Arms: Group A
Device: Shoulder implant — Reverse shoulder arthroplasty device

SUMMARY:
The study is a prospective, multi-center, randomized blinded study to determine how repairing the subscapularis vs. not repairing the subscapularis when subjects are implanted with the AltiVate Reverse® Shoulder System for reverse total shoulder arthroplasty affects isometric and isokinetic internal rotational strength. It is hypothesized that patients in which the subscapularis is repaired will have improved postoperative isometric and isokinetic internal rotational strength.

DETAILED DESCRIPTION:
Reverse shoulder arthroplasty (RSA) is performed to provide improvement in pain relief and restoration of function in patients with rotator cuff tear arthropathy and massive irreparable rotator cuff tears . Traditional total shoulder designs failed to address the unique mechanics of shoulders with deficient rotator cuffs. Different prosthesis designs exist for RSA, all of which increase the deltoid lever arm to provide a stable fulcrum for active elevation in a rotator cuff deficient shoulder.

The Reverse® Shoulder Prosthesis (RSP®) (DJO Surgical) sought to address issues correlated to the Grammont design by lateralizing the center of rotation as well as utilizing a central compressive screw with a 5.0-mm peripheral locking screws for fixation and a glenosphere .

Despite the success of the lateralized design, the effect of the repair of the subscapularis tendon during RSA on shoulder strength, range of motion, and shoulder function remains inconclusive. The rationale for repairing the subscapularis during RSA include anatomic preservation of a functioning rotator cuff muscle, an increased potential for internal rotation, better joint protection, and more stability. The reasoning for not repairing the subscapularis include that it may be biomechanically unfavorable for both the deltoid and the posterior rotator cuff, limiting the range of motion.

As such, this randomized study aims to address if subscapularis repair impacts isometric and isokinetic internal rotational strength, with shoulder function and complications as secondary objectives, when patients are implanted with the AltiVate Reverse® device.

The study will take place at multiple sites across the United States and will be managed by the DJO Surgical Clinical Affairs Department.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥21 years of age
2. Subject is scheduled for reverse shoulder arthroplasty with the AltiVate Reverse device due to primary diagnosis of severe arthropathy with a grossly deficient rotator cuff
3. Subject's sub scapularis has been determined from MRI to be sufficient to repair
4. Subject is willing and able to comply with the study schedule and assessments
5. Subject is likely to be available for evaluation for the duration of the study
6. Subject is willing and able to sign the informed consent

Exclusion Criteria:

1. Subject is indicated for reverse shoulder arthroplasty for other indications (revision arthroplasty, proximal humerus fracture, etc.), addition of latissimus transfer or pectoralis major transfer
2. Subject has metal allergies or sensitivity
3. Subject has an active infection at or near the site of implantation
4. Subject has a nonfunctional deltoid muscle
5. Subject has neuromuscular compromise condition of the shoulder
6. Subject has known active metastatic or neoplastic diseases, Paget's disease or Charcot's disease
7. Subject is currently on or planning to be on chemotherapy or radiation
8. Subject has had chemotherapy or radiation within the last 6 months
9. Subject is currently taking > 5mg/day corticosteroids (e.g. prednisone), excluding inhalers, within 3 months prior to surgery
10. Female subjects who are pregnant or planning to become pregnant within the study period
11. In the investigator's opinion, the subject is unable to understand the study or be compliant with the follow up or has a history of non-compliance with medical advice
12. Subject has a history of any cognitive or mental health status that would interfere with study participation
13. Subject is abusing alcohol or drugs or is undergoing active treatment for substance abuse (e.g., recreational drugs, narcotics, or alcohol).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in isometric and isokinetic internal rotational strength of abductors | 6 months, and 1, 2, 5 and 10 years
  Maximal isometric strength of shoulder abductors and measured in kilograms using a force gauge
Change in isometric and isokinetic internal rotational strength of flexors | 6 months, and 1, 2, 5 and 10 years
  Maximal isometric strength of shoulder flexors measured in kilograms using a force gauge
Change in isometric and isokinetic internal rotational strength of internal rotators | 6 months, and 1, 2, 5 and 10 years
  Maximal isometric strength of shoulder measured internal rotators in kilograms using a force gauge
Change in isometric and isokinetic internal rotational strength of external rotators | 6 months, and 1, 2, 5 and 10 years
  Maximal isometric strength of shoulder measured external rotators in kilograms using a force gauge

SECONDARY OUTCOMES:
To evaluate change in shoulder ROM with the AltiVate Reverse® Shoulder | 6 months, and 1, 2, 5 and 10 years
  Examine operative shoulder active forward elevation
To evaluate change in shoulder ROM with the AltiVate Reverse® Shoulder | 6 months, and 1, 2, 5 and 10 years
  Examine operative shoulder active abduction
To evaluate change in shoulder ROM with the AltiVate Reverse® Shoulder | 6 months, and 1, 2, 5 and 10 years
  Examine operative shoulder active external rotation
To evaluate change in shoulder ROM with the AltiVate Reverse® Shoulder | 6 months, and 1, 2, 5 and 10 years
  Examine operative shoulder active internal rotation
To evaluate change in shoulder functionality with the AltiVate Reverse® Shoulder | 6 weeks,6 months, and 1, 2, 5 and 10 years
  Examine change in ASES score
To evaluate change in shoulder functionality with the AltiVate Reverse® Shoulder | 6 weeks, 6 months, and 1, 2, 5 and 10 years
  Examine change in pain per ASES assessment
To evaluate change in shoulder functionality with the AltiVate Reverse® Shoulder | 6 weeks,6 months, and 1, 2, 5 and 10 years
  Examine change in SST score
To evaluate change in general health with the AltiVate Reverse® Shoulder | 6 weeks, 6 months, and 1, 2, 5 and 10 years
  Examine change in VR-12
To evaluate change in the radiographs of AltiVate Reverse® Shoulder | 6 weeks, 6 months, and 1, 2, 5 and 10 years
  Examine radiographic parameters
To evaluate device survivorship of the AltiVate Reverse® Shoulder | 6 weeks, 6 months, and 1, 2, 5 and 10 years
  Examine adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Knowlton, MS, CRA, Study Director — DJO Global
Locations (4):
- United States (4):
  - St. Luke's Hospital, St Louis, Missouri
  - NYU Langone Center for Musculoskeletal Care, New York, New York
  - Rothman Institute, Philadelphia, Pennsylvania
  - Texas Orthopedic Group, Houston, Texas

IPD SHARING:
Plan to Share IPD: No